CLINICAL TRIAL: NCT06847685
Title: Mechanisms of Uterine Fluid Absorption During Early Pregnancy
Brief Title: Mechanisms of Uterine Fluid Absorption During Early Pregnancy ( ELF Study)
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00423161; R01HD114750 (NIH)
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Endometriosis; Endometrioma
Keywords: Endometriosis; Endometrial biopsy
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endometrial biopsy samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women between the ages of 18 and 45 years with or without endometriosis: 50 women with endometriosis (cases) and 50 without endometriosis (controls)
- Women between the ages of 18 and 45 years with or without endometrial cavity fluid undergoing IVF: 20 women with endometrial lumen fluid and 20 women without endometrial lumen fluid

SUMMARY:
The researchers are evaluating mechanisms of uterine fluid absorption during early pregnancy

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be a healthy woman between the ages of 18 and 45 years.
2. Women with diagnosed endometriosis or infertility (cases).
3. Women without a diagnosis of endometriosis or infertility (controls).
4. Subject must have regular menstrual cycles.
5. Subject must have a body mass index (BMI) between 18 and 40.
6. Subject must be or have been sexually active or have had a previous vaginal exam that used a speculum.
7. Subject must be able to understand and provide consent to procedures and use/disclosure of protected health information.
8. No history of Chlamydia trachomatis, Mycoplasma genitalium, Neisseria gonorrhoeae, hepatitis B, and HIV.
9. For IVF study subjects, a minimum endometrial thickness of 7mm at the time of sample collection.

Exclusion Criteria:

1. Pregnant women.
2. Study subjects with endometrial cancer.
3. Study subjects with a history of endometrial ablation.
4. Study subjects with undiagnosed uterine bleeding.
5. Women with reproductive diseases that affect the endometrium (such as fibroids or uterine polyps that distort endometrial cavity).
6. Study subjects with an intrauterine device (IUD).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women between the ages of 18-45 with or without endometriosis.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Expression levels of selected ion channels in human endometrium biopsies across the menstrual cycle. | 5 years
  Immunolocalization of ion channel levels ENaCα, SLC5A1 and SLC5A3 in endometrial tissues.

SECONDARY OUTCOMES:
Compare relative protein expression of ENaCα, SLC5A1 and SLC5A3 by immunohistochemistry | 5 years
  Compare relative protein expression of ENaCα, SLC5A1 and SLC5A3 by immunohistochemistry in the human endometrial biopsies from women with or without endometriosis.

CONTACTS AND LOCATIONS:
Overall Officials: James Segars, MD, Study Chair — Johns Hopkins University; Bhuchitra Singh, MD, MPH, MS, MBA, Study Director — Johns Hopkins University
Locations (3):
- United States (3):
  - University of Georgia, Athens, Georgia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Rutgers University, Piscataway, New Jersey

IPD SHARING:
Plan to Share IPD: No